CLINICAL TRIAL: NCT06092515
Title: EZAFFAW - Efficacy of Zinc Fortified Fermented Wheat Flour: Randomized Controlled Trial
Brief Title: Efficacy of Zinc Fortified Fermented Wheat Flour
Acronym: EZAFFAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Bahauddin Zakariya University (Other); University of California (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Dr Jai Kumar Das, Assistant Professor and Assistant Director, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-8164-23704
Record Dates: First submitted 2023-09-22; First posted 2023-10-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Malnutrition; Diabetes; Inflammation; Conjunctivitis
Keywords: Zinc; Fortification; Micronutrient; Flour; Trial; Deficiencies
MeSH Terms: conditions — Malnutrition; Diabetes Mellitus; Inflammation; Conjunctivitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: This clinical trial investigates the health impact of consuming various types of wheat flour flatbreads among adolescent and adult females. The primary focus is on assessing zinc status and metabolic health in individuals at high risk of zinc deficiency and Type 2 Diabetes (T2DM). The study encompasses both fermented and unfermented flatbreads made from wheat variants with different zinc content and "post-harvest fortified wheat flour.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This clinical trial will be conducted with a double-blind design
  Participant Blinding:
  Participants will not be informed about which specific type of flatbread they are receiving. Each participant will receive their assigned flatbread without knowledge of whether it falls into the fermented high zinc, unfermented high zinc, post-harvest fortified, or low zinc category.
  Investigator and outcomes assessor Blinding:
  The investigators and research staff responsible for data collection and assessment will also be unaware of the treatment assignments. They will not be involved in the preparation of the flatbreads to ensure that their observations and assessments are unbiased.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fermented High Zinc Wheat Flour Flatbread (Experimental): Participants in this arm will receive fermented whole wheat flatbreads made from wheat variants with a high zinc content, ranging. These flatbreads are prepared through traditional fermentation methods.
  Interventions: Dietary Supplement: Fermented High Zinc Wheat Flour Flatbread
- Unfermented High Zinc Wheat Flour Flatbread (Experimental): Participants in this arm will receive unfermented whole wheat flatbreads made from wheat variants with a high zinc content. These flatbreads provide a source of bioavailable zinc without the fermentation process.
  Interventions: Dietary Supplement: Unfermented High Zinc Wheat Flour Flatbread
- Fortified Wheat Flour flatbread (Experimental): Participants in this arm will receive flatbreads made from whole wheat flour fortified post-harvest to contain a zinc content
  Interventions: Dietary Supplement: Post-Harvest Fortified Whole Wheat Flour Flatbread
- Low Zinc Wheat flatbread (Active Comparator): Participants in this arm will receive whole wheat flatbreads made from wheat variants with a low zinc content
  Interventions: Dietary Supplement: Low Zinc Whole Wheat Flour Flatbread (Control Group)

INTERVENTIONS:
Dietary Supplement: Fermented High Zinc Wheat Flour Flatbread — * Participants in this group will receive flatbreads made from fermented high zinc wheat flour.
  * The flatbreads will be prepared using traditional fermentation methods.
  * These flatbreads will be provided to participants to consume daily, along with vegetables or pulses (daal), for six days a week over the course of six months.
  Arms: Fermented High Zinc Wheat Flour Flatbread
Dietary Supplement: Unfermented High Zinc Wheat Flour Flatbread — * Participants in this group will receive flatbreads made from unfermented high zinc wheat flour,
  * The flatbreads will not undergo a fermentation process.
  * These flatbreads will be provided to participants to consume daily, along with vegetables or pulses (daal), for six days a week over the course of six months.
  Arms: Unfermented High Zinc Wheat Flour Flatbread
Dietary Supplement: Post-Harvest Fortified Whole Wheat Flour Flatbread — * Participants in this group will receive flatbreads made from whole wheat flour fortified post-harvest
  * These fortified flatbreads will be provided to participants for daily consumption, along with vegetables or pulses (daal), for six days a week over the course of six months.
  Arms: Fortified Wheat Flour flatbread
Dietary Supplement: Low Zinc Whole Wheat Flour Flatbread (Control Group) — * Participants in this group will serve as the control group.
  * They will receive flatbreads made from whole wheat flour with a low zinc content
  * These low zinc flatbreads will be provided to participants for daily consumption, along with vegetables or pulses (daal), for six days a week over the course of six months. six days a week over the course of six months.
  Arms: Low Zinc Wheat flatbread

SUMMARY:
Zinc is a pivotal micronutrient that participates in numerous essential metabolic pathways within the human body. Its multifaceted role makes the manifestations of zinc deficiency remarkably nonspecific and age-dependent. In children, zinc deficiency can manifest as growth retardation, cognitive impairment, recurrent infections, and other diverse symptoms. Adolescents and adults may experience fertility issues, work capacity impairment, and metabolic disorders due to zinc deficiency. Furthermore, zinc plays a crucial role in maintaining immune function, particularly in the elderly, where recurrent infections can be a notable outcome of deficiency. Given its fundamental importance, the potential benefits of zinc supplementation and fortification strategies have been explored, with some evidence indicating positive effects on health outcomes such as childhood mortality, diarrhea morbidity, and even risk factors for conditions like Type 2 Diabetes (T2DM) and cardiovascular disease (CVD). Understanding zinc's significance in these metabolic processes is vital for addressing deficiencies and improving public health.

A study is needed to assess the effect of various types of fermented and unfermented wheat flour flatbread and its impact on health including zinc status, anthropometric outcomes, risk of T2DM and CVD and morbidity on adolescent and adult females. The whole wheat flatbread trial would be ideal to inform policy as it is regularly consumed in Sindh as most people rely on chakki for wheat grinding and it is used commonly to make roti at home.

DETAILED DESCRIPTION:
STUDY DESIGN

This will be an individually randomized, double-blind efficacy trial in Mithi, District Tharparkar, Sindh, Pakistan. This district is among the most impoverished in Sindh, characterized by a tropical desert climate with extremely hot mornings. Approximately 87% of the population in Tharparkar lives below the poverty line. Due to its challenging demographics and environmental conditions, the region has endured severe droughts and faces the highest level of food insecurity among Sindh districts. It is concerning that 60% of children under five years suffer from stunting, 33.3% from wasting, and nearly 19.8% experience both conditions simultaneously. Additionally, approximately 40.4% of non-pregnant women of reproductive age are underweight. Tharparkar has been selected for this study due to its alarming rates of malnutrition and micronutrient deficiencies, making it an ideal location to assess the effectiveness of fortified wheat flour.

RESEARCH QUESTION

* Primary Does consumption of whole wheat flatbread made with fermented and unfermented 'high zinc wheat' or with 'post-harvest zinc-fortified wheat flour' improve zinc status and metabolic health among adolescents (10-19 years) and adult women (20-40 years) at high risk of zinc deficiency and T2DM compared to 'low zinc' whole wheat flatbread?
* Secondary Does an increase in bioavailable dietary zinc intake improve indicators for predicting the risk of T2DM in adolescents and adult women at high risk of zinc deficiency? SPECIFIC OBJECTIVES
* Primary To evaluate the efficacy of whole wheat flatbread made with fermented and unfermented 'high zinc wheat' or post-harvest zinc-fortified wheat on zinc status/zinc deficiency and metabolic health among adolescents and adult women at high risk of zinc deficiency when compared to the 'low zinc' whole wheat flatbread.
* Secondary To assess if an increase in bioavailable dietary zinc intake improves indicators for predicting the risk of T2DM in adolescents and adult women at high risk of zinc deficiency.

PARTICIPANTS The study will include adolescents (10-19 years) and adult women (20-40 years) INTERVENTION

Participants will be randomly divided into four groups according to the four-arm design in a 1:1:1:1 ratio. A total of 1000 participants would be randomly allocated to each of the groups in a 1:1:1:1 ratio.

* Group 1: will receive fermented high zinc wheat flour flatbread
* Group 2: will receive unfermented high zinc wheat flour flatbread
* Group 3: will receive fortified (post-harvest) whole wheat flour flatbread
* Group 4: will receive low zinc whole wheat flour flatbread

It would be a six-month intervention, where the participants would be given flatbread with a vegetable/pulse (daal) each day for six days a week for six months. On average, 2-3 flatbreads will be provided per participant (this was ascertained in the pilot activity). This would be provided at the school/college campus at lunch time i.e., at 1.30pm and all the participants enrolled in the study would be directly observed each day for the amount consumed and adult women would be provided meal at a community place.

OUTCOMES

Primary:

* Serum zinc concentration
* Zinc deficiency
* HbA1C
* Fasting blood glucose
* Insulin levels
* HOMA-IR (cut-off >2) (27)
* Lipid profile (total cholesterol, very low-density lipoprotein (VLDL), low-density lipoprotein (LDL), high-density lipoprotein (HDL); triglycerides (TGs))
* Red blood cell membrane fatty acids concentrations

Secondary:

* Anthropometric measurements:

  * Height
  * Weight
  * Mid upper arm circumference (MUAC)
  * Waist circumference
* Body Mass Index (BMI) - Severe thinness, thinness, normal weight, overweight, obese
* Blood Pressure
* Anemia
* School attendance/ performance
* Dietary intakes through 24hr dietary recall.
* Morbidity - Diarrhea, Acute respiratory infection (ARI) etc.

Compliance:

* Number of days each participant had flatbread
* Flatbread consumed (weight) each day

SAMPLE SIZE CALCULATION The study sample size was calculated based on an individually randomized four arm design on the primary outcome of mean serum zinc levels and HbA1c. The mean HbA1c taken was 5.62% (SD 1.96) and mean zinc was 79.5 µg/dL (SD 35.9) according to NNS-2018. The serum zinc data for the Tharparkar district was taken from NNS 2018, while there is no data on area specific estimates for T2DM and HbA1c. A recent national community-based survey conducted in 2019 found that the prevalence of diabetes (19.09%) and pre-diabetes (12.79%) in rural areas of Pakistan is high compared to the urban areas of Pakistan (diabetes: 15.75%; prediabetes: 9.89%) and the overall mean HbA1c was 5.62% (SD 1.96).

The sample size was calculated with a power of 0.8 and alpha of 0.05 to detect a difference of at least 0.12 effect size in the mean serum zinc levels between groups and to detect a 0.2 effect size in the mean HbA1c levels with a dropout rate of 10%.

The sample size calculated is 250 participants. A total of 1000 participants would be randomly allocated to each of the groups in a 1:1:1:1 ratio.

Baseline, midline, and end-line data collection.

All the participants will be assessed at baseline, and at endline. Data will be collected on socio-demographic factors, dietary intake through 24-hour dietary recall, anthropometry (weight, height, MUAC, waist circumference), blood pressures and blood samples for bio-chemical analysis including serum zinc levels, FBS, HbA1C, insulin at both baseline and endline, while lipid profile and RBC membrane fatty acids would be done at endline only. At midline, 24-hour dietary recalls, serum zinc, and HbA1C will be taken on a subset from each group. For morbidity and ARI, a two-week data collection will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents aged 10-19 years
* Adult women aged 20-40 years.
* Wheat as a staple part of their diet

Exclusion Criteria:

* Severe Malnutrition
* Pregnant or Lactating
* Chronic Diseases
* Participation in Similar Programs
* Individuals taking vitamin or mineral supplements at the time of enrollment
* Planned Relocation from the study area within the next 6-7

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1044 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Zinc Status | Baseline and six months post intervention
  The primary outcome is the measurement of serum zinc status (micrograms per deciliter (μg/dL) in participants. This includes assessing the concentration of zinc in serum samples. Changes in serum zinc levels will be compared between the four intervention groups.
Fasting Blood Glucose | Baseline and six months post-intervention.
  This outcome assesses changes in participants' fasting blood glucose levels, measured in milligrams per deciliter (mg/dL). It aims to understand alterations in blood glucose levels resulting from flatbread interventions.
HbA1C Levels | Baseline and six months post-intervention.
  This measure evaluates HbA1C levels, expressed as a percentage (%). It provides insights into long-term blood glucose control, helping assess the impact of dietary interventions.
Insulin Levels | Baseline and six months post-intervention.
  This measure assesses participants' insulin levels, measured in microunits per milliliter (μU/mL). It helps in understanding changes in insulin sensitivity as a result of dietary interventions.
Lipid Profiles | Six months post-intervention.
  This measure assesses participants' lipid profiles, with the unit of measure to be specified (e.g., milligrams per deciliter, mg/dL). It provides insights into changes in lipid levels and their potential effects on overall body composition due to dietary interventions.
Zinc Deficiency (%) | Baseline and six months post intervention
  This primary outcome evaluates the prevalence of zinc deficiency among participants and it would be compared across the four groups.
Red blood cell membrane fatty acids concentrations | At six months post intervention
  This outcome measures the red blood cell membrane fatty acids concentrations as a percentage (%) and This would be compared across the four groups.

SECONDARY OUTCOMES:
Change in Weight (kg) | Six months post intervention
  This outcome assesses changes in participants' weight, measured in kilograms (kg), to understand alterations in their physical characteristics resulting from flatbread interventions.
Change in Height (m) | Six months post intervention
  This measure evaluates changes in participants' height, measured in meters (m), to determine any variations in their physical stature due to dietary changes.
Change in BMI (kg/m²) | Six months post intervention
  Body Mass Index (BMI) is calculated using weight (in kilograms) and height (in meters) and is measured in kg/m². This measure provides insights into participants' overall body composition and potential effects of dietary changes.
Acceptability and Adherence Assessment | Six months post intervention
  Secondary outcomes focus on participants' satisfaction and adherence to dietary interventions, offering insights into the feasibility and acceptability of the intervention.
School Attendance and Academic Performance | Six months post intervention
  This outcome aims to determine if the intervention resulted in better school attendance and academic performance (determined by school) among participants.
Morbidity | Six months post intervention
  This outcome monitors the incidence of common health infections as diarrhea and acute respiratory infections and will be reported as a percentage (%).
Anemia | Six months post intervention
  Anemia will be assessed through hemoglobin levels and will be reported as a percentage (%). This will determine whether there was a difference among the four groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jai K Das, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Das JK, Padhani ZA, Khan M, Mirani M, Rizvi A, Chauhadry IA, Yasin R, Ismail T, Akhtar S, Begum K, Iqbal J, Humayun K, Naseem HA, Malik KA, Bhutta ZA. Efficacy of Zinc Fortified and Fermented Wheat Flour (EZAFFAW): A randomized controlled trial protocol. PLoS One. 2024 Jun 20;19(6):e0304462. doi: 10.1371/journal.pone.0304462. eCollection 2024. PMID 38900773